CLINICAL TRIAL: NCT06833463
Title: Tacrolimus and Risk Factors for Glucose Metabolism Disorders in Kidney Transplant Patients
Acronym: TARGET
Status: Recruiting | Type: Observational
Sponsor: Chiesi Poland Sp. z o.o. (Industry)
Responsible Party: Sponsor
Other Study IDs: CHI-PL-ENV-03
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Kidney Transplant
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: LCP Tacro (tacrolimus) — Treatment with LCP Tacro will begin on the day of the kidney transplant. If a patient is switching from another form of tacrolimus to LCP Tacro, the transition will be completed no later than day 8, following the standard procedures of the medical institution.

SUMMARY:
Many people who receive a kidney transplant develop problems with how their body processes sugar (glucose). This includes conditions like prediabetes and diabetes, which can lead to more health issues, such as heart problems and infections.

One of the main medications used after a kidney transplant, called tacrolimus, can contribute to these sugar problems. Tacrolimus helps protect the new kidney, but it can also harm the cells in the pancreas that produce insulin, a hormone that controls blood sugar. Other factors, such as stress on the body and insulin resistance, can make things worse.

The effect of tacrolimus on blood sugar may depend on how the body processes the drug. Some people break down tacrolimus quickly (fast metabolizers), so they need higher doses to reach the right level in their blood. Others break it down more slowly (slow metabolizers) and require lower doses. Doctors can measure how fast someone metabolizes tacrolimus using aparameter called the concentration-to-dose (C/D) ratio.

This study aims to find out what increases the risk of developing blood sugar problems after a kidney transplant. It will focus on how quickly patients process tacrolimus and whether this affects their risk of developing diabetes. The study will also look at how common these issues are in kidney transplant patients in Poland.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Recipients of a kidney transplant from a living or deceased donor
* Standard immunosuppressive regimen post-kidney transplantation (KTx) including Envarsus®
* LCP Tacrolimus therapy initiated from the day of KTx or conversion from another tacrolimus formulation to LCP Tacrolimus by day 8 at the latest, according to the institution's routine practice
* Informed patient consent to participate in the study

Exclusion Criteria:

* Diagnosis of diabetes (type 1 or type 2) treated with diet or glucose-lowering drugs
* Random glycemia/HbA1c levels justifying a diagnosis of diabetes at the time of study enrollment
* Kidney retransplantation
* Recipients of a multi-organ transplant
* Use of glucagon-like peptide-1 (GLP-1) receptor agonists for weight loss
* Use of flozins for renal or cardiac indications
* Chronic use of drugs affecting carbohydrate metabolism, such as glucocorticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult kidney graft receipients transplanted in the participating study sites
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Glucose metabolism disorders during tacrolimus treatment | The endpoint will be determined at 3, 6, and 12 months after transplantation
  Percentage of patients diagnosed with:
  * Impaired fasting glucose and/or glucose intolerance (prediabetes)
  * Post-transplant diabetes mellitus (PTDM) requiring pharmacotherapy,
Risk factors for glucose metabolism disorders | 3, 6, and 12 months after transplantation
  Odds ratio for glucose metabolism disorders (prediabetes, PTDM) for the following variables: the rate of tacrolimus metabolism, cumulative tacrolimus exposure, cumulative glicocorticosteroid exposure, age, sex, body mass index

SECONDARY OUTCOMES:
Fasting glucose | over a period of 1-12 months
  Changes in mean fasting glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Alicja Dębska-Ślizień, Professor, Principal Investigator — Department of Nephrology, Transplantology and Internal Diseases, Medical University of Gdansk, Gdansk, Poland
Locations (6):
- Poland (6):
  - Department of Nephrology, Transplantology and Internal Diseases, Medical University of Gdansk, Gdansk
  - Clinical Department of Nephrology, Dialysis, Transplantology and Internal Medicine, Krakow
  - Department of Internal Diseases and Transplant Nephrology, Medical University of Lodz, Lodz
  - Department of Transplantology and General Surgery, Provincial Hospital, Poznan
  - Department and Clinic of Nephrology, Dialysis and Internal Medicine, Medical University of Warsaw, Warsaw
  - Department and Clinic of Nephrology and Transplantation Medicine, University Clinical Hospital, Wroclaw

IPD SHARING:
Plan to Share IPD: Undecided